CLINICAL TRIAL: NCT06807801
Title: BIDAP - Baby Swim As an Intervention for Depressive Symptoms and Lacking Attachment During the Postpartum Period
Brief Title: Baby Swim As an Intervention for Depressive Symptoms and Lacking Attachment During the Postpartum Period
Acronym: BIDAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIDAP
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Depression - Major Depressive Disorder; Attachment; Postpartum
Keywords: depression; attachment; postpartum; baby swimming
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: The project is an interventional study in the form of an RCT with a waitlist control group and will be conducted at Uppsala University Hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Waiting list (Active Comparator): After completing the baseline questionnaire at T0, participants will be randomized into two groups: half will receive the intervention immediately (the treatment group), while the other half will receive it after seven months (the waitlist control group).
  Interventions: Behavioral: Baby swimming
- Intervention (Active Comparator): Participants in the treatment group will be contacted by a researcher and invited to an introductory meeting at the swimming facility, where they will receive information about the baby swimming course from the instructor. The course will take place twice a week for five weeks, totaling 10 sessions of 30 minutes each. During the sessions, mothers will be encouraged to engage in physical contact, maintain eye contact, and respond to their baby's signals. The course will also include water safety exercises.
  Interventions: Behavioral: Baby swimming

INTERVENTIONS:
Behavioral: Baby swimming — Participants in the treatment group will be contacted by a researcher and invited to an introductory meeting at the swimming facility, where they will receive information about the baby swimming course from the instructor. The course will take place twice a week for five weeks, totaling 10 sessions of 30 minutes each. During the sessions, mothers will be encouraged to engage in physical contact, maintain eye contact, and respond to their baby's signals. The course will also include water safety exercises.

SUMMARY:
Mental health issues are very common during and after pregnancy, and studies from around the world indicate that 10-15% of all pregnant and postpartum women experience depression. Risk factors for developing depression include a history of depression, low levels of social support, and stressful life events. The symptoms are the same as for depression during other periods of life, but often include feelings of inadequacy regarding motherhood, along with associated feelings of shame or guilt. Obsessive thoughts directed toward the baby may also be part of the symptomatology. Such thoughts are typically experienced as frightening by the mother but, in the vast majority of cases, do not pose any risk to the child. Maternal depression can also affect a mother's ability to bond with her baby, and difficulties in forming an attachment can, in turn, increase and perpetuate depressive symptoms. In the long term, insecure attachment between mother and child can lead to behavioral problems in the child, such as aggression and avoidance, anxiety and depression in adolescence, negative effects on cognitive development, and trust issues in close relationships.

Baby swimming is a structured form of interaction that takes place in 34-degree Celsius water in a calm environment, aiming to teach the baby vital skills while stimulating social, intellectual, and motor development. At least one parent actively participates and is encouraged to perform various exercises. These activities strengthen the bond between the baby and the parent and contribute to making time in the water a safe and enjoyable experience. Previous studies have shown that baby swimming can improve attachment between parent and child.

In the present project, the aim is to investigate whether baby swimming can be used as an intervention for depressive symptoms in new mothers and whether this intervention can reduce depressive symptoms while also strengthening the bond between mother and child.

ELIGIBILITY:
Inclusion Criteria:

Women who have

* given birth at full term
* are 18 years or older
* have a baby aged 3-7 months at the time of inclusion
* exhibit depressive symptoms according to the EPDS scale.

Exclusion Criteria:

* Multiple pregnancy (twins, triplets)
* Known psychotic disorder or bipolar disorder
* Inability to communicate adequately in Swedish or English, or inability to read and complete digital questionnaires in Swedish or English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms | Seven months follow up
  Self-reported depressive symptoms measured by the Edinburgh Postnatal Depression Scale

SECONDARY OUTCOMES:
Attachment | Seven months follow up
  Measured by the Postpartum Bonding Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Uppsala University, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Undecided